CLINICAL TRIAL: NCT03000868
Title: Comparison of Small Colorectal Polyp Removal Using Cold Endoscopic Mucosal Resection With Hot Endoscopic Mucosal Resection: a Pilot Study
Brief Title: Comparison of Small Colorectal Polyp Removal Using Cold EMR With Hot EMR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled.
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Chang Hwan Park, Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNUH-2016-252
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Colonic Polyps
Keywords: Colonic Polyps; Endoscopic Mucosal Resection; Colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cold EMR group (Experimental): Patients who have small colorectal polyps (<1cm) who receive endoscopic mucosal resection using snare without electrocautery.
  Interventions: Procedure: Cold endoscopic mucosal resection
- Hot EMR group (Active Comparator): Patients who have small colorectal polyps (<1cm) who receive endoscopic mucosal resection using snare with the use of electrocautery.
  Interventions: Procedure: Hot endoscopic mucosal resection

INTERVENTIONS:
Procedure: Cold endoscopic mucosal resection — Cold endoscopic mucosal resection (EMR) means removing small colorectal polyps (<1cm) with snare without the use of electocautery after injection of normal saline into the submucosa.
  Arms: Cold EMR group
Procedure: Hot endoscopic mucosal resection — Hot endoscopic mucosal resection (EMR) means removing small colorectalpolyps (<1cm) with snare without the use of electocautery after injection of normal saline into the submucosa.
  Arms: Hot EMR group

SUMMARY:
This study evaluates the efficacy of small colorectal polyp removal using cold endoscopic mucosal resection with hot endoscopic mucosal resection. Half of the participants will receive cold endoscopic mucosal resection, while the other half will receive hot endoscopic mucosal resection.

DETAILED DESCRIPTION:
Colorectal polyps are considered as precancerous lesions and endoscopical resection is currently the treatment of choice when it is possible.

Colorectal polyps are classified into diminutive polyps (<5mm in diameter), small polyps (6-9mm in diameter), and large polyps (>1cm in diameter). There are several endoscopical treatment methods: cold biopsy forceps polypectomy, cold snare polypectomy, hot biopsy forceps polypectomy, hot snare polypectomy, and endoscopic mucosal resection. Cold polypectomy means mechanical removal of the polyp with snare or biopsy forceps without the use of electrocautery, and hot polypectomy means removal of the polyp with the use of electocautery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal polyps that are <1cm in diameter who need endoscopic mucosal resection.

  * Patients who gave informed consents to this study.

Exclusion Criteria:

* Patients under the age of 19
* Patients who are receiving antiplatelet or anticoagulant therapies
* Patients with hypercoagulability (i.e., liver cirrhosis, hemophilia, end-stage renal disease, or chronic kidney disease)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Complete removal of the colorectal polyp | At the time of the procedure (endoscopic mucosal resection)
  The resected specimen will be reviewed microscopically to assess complete resection including the lateral and base margins

SECONDARY OUTCOMES:
Procedure time | At the time of the procedure (endoscopic mucosal resection)
  The time needed for the hot EMR vs cold EMR (minutes) will be assessed.
Complication after endoscopic mucosal resection | Within 1 month
  Procedure-related complications (bleeding, perforation, and post-coagulation syndrome) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-hwan Park, M.D., Ph.D, Study Director — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not planned to be shared to other researchers.

REFERENCES:
- [Background] Horiuchi A, Makino T, Ichise Y, Kajiyama M, Kato N, Tanaka N. Comparison of newly found polyps after removal of small colorectal polyps with cold or hot snare polypectomy. Acta Gastroenterol Belg. 2015 Dec;78(4):406-10. PMID 26712051
- [Background] Lee SH, Shin SJ, Park DI, Kim SE, Hong SP, Hong SN, Yang DH, Lee BI, Kim YH, Kim HS, Yang SK, Kim HJ, Kim SH, Kim HJ; Multi-Society Task Force for Development of Guidelines for Colorectal Polyp Screening, Surveillance and Management. [Korean guidelines for colonoscopic polypectomy]. Korean J Gastroenterol. 2012 Feb;59(2):85-98. doi: 10.4166/kjg.2012.59.2.85. Korean. PMID 22387834
- [Background] Horiuchi A, Nakayama Y, Kajiyama M, Tanaka N, Sano K, Graham DY. Removal of small colorectal polyps in anticoagulated patients: a prospective randomized comparison of cold snare and conventional polypectomy. Gastrointest Endosc. 2014 Mar;79(3):417-23. doi: 10.1016/j.gie.2013.08.040. Epub 2013 Oct 11. PMID 24125514